CLINICAL TRIAL: NCT02229487
Title: The Relationship Between Sleep and Glucose Tolerance in Prediabetes: the Role of GLP-1 in Short Sleepers
Acronym: Sleep GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sirimon Reutrakul, Associate Professor, Ramathibodi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-57-16
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-09

CONDITIONS: Prediabetes
Keywords: Prediabetes; Short sleepers; GLP-1
MeSH Terms: conditions — Prediabetic State | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Sleepers (Active Comparator): Prediabetes patients with normal sleep duration (7-8 hours/ night) as measured objectively
  Interventions: Other: Oral glucose tolerance
- Short Sleepers (Experimental): Prediabetes patients with short sleep duration (<6 hours/night) as measured objectively
  Interventions: Other: Oral glucose tolerance

INTERVENTIONS:
Other: Oral glucose tolerance

SUMMARY:
Hypothesis

1. Prediabetes patients who have insufficient sleep will have worse glucose tolerance than those with normal sleep duration.
2. Prediabetes patients with short sleep will have a delayed or reduced GLP-1 response to a standardized meal

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prediabetes (HbA1c 5.7-6.4% or history of fasting plasma glucose 100-125 mg/dl) who receive medical care at Ramathibodi Hospital
2. Age 18 or older
3. Can understand Thai (speaking, listening and reading)
4. Agree to participate by written informed consent

Exclusion Criteria:

1. Those who depend on others for feeding (such as stroke patients)
2. Shift workers
3. History of congestive heart failure or low ejection fraction
4. Chronic obstructive pulmonary disease, end stage renal disease or chronic liver disease (AST or ALT > 3 times the upper limit of normal)
5. Use of medications: opioids/ narcotics , alpha blockers (prazosin, doxazosin, terazosin), clonidine, methyldopa, nitroglycerin
6. Patients with permanent pacemaker
7. History of previous stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Sleepers: Prediabetes patients with normal sleep duration (>=6.5 hours/ night) as measured objectively
  Oral glucose tolerance
- Short Sleepers: Prediabetes patients with short sleep duration (=<5.75 hours/night) as measured objectively
  Oral glucose tolerance
Period: Overall Study
Arm/Group | Normal Sleepers | Short Sleepers
Started | 24 | 27
Completed | 24 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Sleeper: Sleep duration as measured by actigraphy >=6.5 h/night
- Short Sleeper: Sleep duration as measured by actigraphy =<5.75 h/night
- Total: Total of all reporting groups
Arm/Group | Normal Sleeper | Short Sleeper | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.8) | 55.8 (6.7) | 55.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Thai | 24 | 27 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 24 | 27 | 51
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (3.2) | 26.8 (3.8) | 26.8 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: GLP-1 Levels in Response to Oral Glucose Tolerance Test
Description: Prediabetes patients with and without short sleep will undergo an oral glucose tolerance test with measurement of GLP-1 levels
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: pmol/l.h
Groups:
- Short Sleepers: Sleep duration as measured by actigraphy =<5.75 h/night
- Normal Sleepers: Sleep duration as measured by actigraphy >=6.5h/night
Arm/Group | Short Sleepers | Normal Sleepers
Number analyzed (Participants) | 27 | 24
pmol/l.h | 16.66 [12.21 to 21.10] | 18.57 [13.42 to 39.15]
Statistical Analysis 1: Comparison: Short Sleepers vs Normal Sleepers; Test type: Other; p = 0.209, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 18 month
Groups:
- Short Sleeper: Sleep duration as measured by actigraphy =<5.7 h/night
Arm/Group | Normal Sleeper | Short Sleeper
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT02229487/Prot_SAP_000.pdf